CLINICAL TRIAL: NCT05948943
Title: A Two-stage Double-blind, Randomized, Placebo-controlled Study to Assess the Efficacy, Safety and Pharmacokinetics of Alpelisib in Pediatric and Adult Patients With Lymphatic Malformations Associated With a PIK3CA Mutation.
Brief Title: Alpelisib in Pediatric and Adult Patients With Lymphatic Malformations Associated With a PIK3CA Mutation.
Acronym: EPIK-L1
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBYL719P12201; 2023-504146-60-00 (Registry Identifier: EU CTIS number)
Record Dates: First submitted 2023-07-04; First posted 2023-07-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lymphatic Malformations
Keywords: Lymphatic malformations (LyM); Cystic lymphangioma; Cystic hygroma; Lymphangioma circumscriptum; Cavernous lymphangioma; Lymphangioma; Macrocystic lymphatic malformation; Microcystic lymphatic malformationn; Alpelisib
MeSH Terms: conditions — Lymphatic Abnormalities; Lymphangioma, Cystic; Lymphangioma | interventions — Alpelisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Adult participants, alpelisib dose 1 (Stage 1) (Experimental): Adult participants (≥18 years of age) who will receive dose 1 of alpelisib an open-label fashion for at least 24 weeks unless they discontinue earlier (Stage 1)
  Interventions: Drug: Alpelisib
- Adult participants, alpelisib dose 2 (Stage 1) (Experimental): Adult participants (≥18 years of age) who will receive dose 2 of alpelisib in an open-label fashion for at least 24 weeks unless they discontinue earlier (Stage 1).
  Interventions: Drug: Alpelisib
- Pediatric participants (6-17 years of age), alpelisib dose 2 (Stage 1) (Experimental): Pediatric participants 6-17 years of age who will receive dose 2 of alpelisib in an open-label fashion for at least 24 weeks unless they discontinue earlier (Stage 1)
  Interventions: Drug: Alpelisib
- Pediatric participants (6-17 years of age), alpelisib dose 3 (Stage 1) (Experimental): Pediatric participants 6-17 years of age who will receive dose 3 of alpelisib in an open-label fashion for at least 24 weeks unless they discontinue earlier (Stage 1).
  Interventions: Drug: Alpelisib
- Adult participants, alpelisib (Stage 2) (Experimental): Adult participants (≥18 years of age) who will receive alpelisib at the dose selected for confirmatory phase in adult participants (Stage 2)
  Interventions: Drug: Alpelisib
- Adult participants, placebo (Stage 2) (Placebo Comparator): Adult participants (≥18 years of age) who will receive matching placebo
  Interventions: Drug: Placebo
- Pediatric participants (6-17 years of age), alpelisib (Stage 2) (Experimental): Pediatric participants (6-17 years of age) who will receive alpelisib at the dose selected for confirmatory phase in pediatric participants (Stage 2)
  Interventions: Drug: Alpelisib
- Pediatric participants (6-17 years of age), placebo (Stage 2) (Placebo Comparator): Pediatric participants (6-17 years of age) who will receive matching placebo
  Interventions: Drug: Placebo
- Pediatric participants (0-5 years of age), alpelisib (Stage 2) (Experimental): Pediatric participants of 0-5 years who will dose 3 of alpelisib in an open-label fashion for at least 24 weeks unless they discontinue earlier
  Interventions: Drug: Alpelisib

INTERVENTIONS:
Drug: Alpelisib — In Stage 1: adult participants (≥18 years of age) will receive dose 1 or dose 2 of alpelisib; pediatric participants (6-17 years of age) will receive dose 2 or dose 3 of alpelisib.
  In Stage 2: Adult participants will receive alpelisib at the dose selected for confirmatory phase in adult participants; pediatric participants (6-17 years of age) will will receive alpelisib at the dose selected for confirmatory phase in pediatric participants; and pediatric participants of 0-5 years of age will receive dose 3 of alpelisib
  Other Names: BYL719
  Arms: Adult participants, alpelisib (Stage 2); Adult participants, alpelisib dose 1 (Stage 1); Adult participants, alpelisib dose 2 (Stage 1); Pediatric participants (0-5 years of age), alpelisib (Stage 2); Pediatric participants (6-17 years of age), alpelisib (Stage 2); Pediatric participants (6-17 years of age), alpelisib dose 2 (Stage 1); Pediatric participants (6-17 years of age), alpelisib dose 3 (Stage 1)
Drug: Placebo — In Stage 2, participants will receive matching placebo for 24 weeks of the study
  Arms: Adult participants, placebo (Stage 2); Pediatric participants (6-17 years of age), placebo (Stage 2)

SUMMARY:
The main purpose of this study in participants with PIK3CA-mutated LyM is to assess the change in radiological response and symptom severity upon treatment with alpelisib film-coated tablets (FCT) as compared to placebo.

DETAILED DESCRIPTION:
This is a phase II/III multi-center study with two stages:

* Stage 1 is designed to select the dose(s) for the confirmatory phase (DSCP) for alpelisib in Stage 2 and will comprise a 24-week open-label core phase in adult (≥18 years of age) and pediatric participants (6-17 years of age) with PIK3CA-mutated LyM, followed by an extension. After eligibility has been confirmed at screening, participants will be randomized in a 1:1 ratio to the different alpelisib doses according to their age. Depending on the results at the end of Stage 1 core phase, the Stage 2 will be opened to adult and/or pediatric participants or the study may be stopped.
* Stage 2 is designed to confirm the efficacy and assess safety of alpelisib at the DSCP in participants with PIK3CA-mutated LyM and will comprise a 24-week randomized, double blind, placebo-controlled confirmatory phase in adult (≥18 years of age) and pediatric participants 6-17 years of age followed by an open-label extension. After eligibility has been confirmed at screening participants will be randomized in a 2:1 ratio to alpelisib or placebo.

Additionally, in parallel, Stage 2 will include a 24-week open-label core phase in pediatric participants 0-5 years of age followed by an extension, if pediatric participants will be enrolling in Stage 2.

Based on the results of the 24-week open-label core phase of Stage 1, the dose(s) for Stage 2 will be selected by Novartis in consultation with the Steering Committee (SC). During the 24-week randomized, double blind, placebo-controlled core phase of Stage 2, an Independent Data Monitoring Committee (DMC) will conduct periodic safety and efficacy reviews to assess the risk benefit profile of the treatment.

ELIGIBILITY:
Key inclusion criteria:

1. Signed informed consent and assent (when applicable) from the participant, parent, legal authorized representative or guardian.
2. Participant must be willing to remain at the clinical site as required by the protocol and be willing to adhere to study restrictions and examination schedules.
3. Participant has a physician confirmed and documented diagnosis of a symptomatic LyM at the time of informed consent (Note: the physician must confirm that the LyM cannot be included under the PROS diagnostic criteria).
4. Participant is not considered as a candidate for or is not willing to receive non-drug therapies including but not limited to sclerotherapy, embolization, and surgery until the completion of Week 24 in Stage 1 and 2.
5. Participant has evidence of a somatic mutation(s) in the PIK3CA gene prior to randomization.
6. Participant has at least one measurable LyM lesion confirmed by BIRC assessment prior to randomization.
7. Participants must be able to ingest study drug (either in tablet form or as a drinkable suspension [Groups 1 to 4] or granules or as an oral suspension [Group 5]) as assessed within 7 days before study treatment start. Drug administration via feeding tubes is allowed.

Key exclusion criteria:

1. Participant has a physician-confirmed and documented diagnosis of PROS at the time of informed consent.
2. Participant has a physician-confirmed and documented diagnosis of a Central Conducting Lymphatic Anomaly, General Lymphatic Anomaly, Gorham-Stout disease, Kaposiform lymphangiomatosis at the time of informed consent.
3. Participant has a known history of Stevens-Johnson syndrome, erythema multiforme, or toxic epidermal necrolysis at the time of informed consent.
4. Participant has an established diagnosis of type I diabetes mellitus or uncontrolled type II diabetes mellitus at the time of informed consent.
5. Participant had previous treatment with alpelisib and/or any other PI3K inhibitors with treatment duration longer than 2 weeks at the time of informed consent.

Other inclusion/exclusion criteria may apply

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2033-05-02 (Estimated)

PRIMARY OUTCOMES:
Stage 2:Radiological response rate at Week 24 of Stage 2 (adult and pediatric (6 - 17 years of age) participants) | Baseline, Week 24
  Radiological response defined by achieving at least 20% reduction in the sum of target lesion volumes (1 to 3 lesions), assessed by MRI by a BIRC at Week 24, provided that none of the individual target lesions has at least 20% increase from baseline and in absence of progression of non-target lesions and without new lesions. The percentage of participants with a radiological response at Week 24 of Stage 2 in adult and pediatric (6-17 years of age) groups will be assessed

SECONDARY OUTCOMES:
Stage 2: Percentage of participants with at least a 1-point improvement compared to baseline based on patient global impression of severity (PGI-S) scale at Week 24 of Stage 2 (adult and pediatric (6 - 17 years of age) participants) | Baseline, Week 24
  PGI-S is a single item measure to assess the overall severity of a patient's condition. This single item instrument uses a 5-point rating scale, which ranges from 1 (no symptoms) to 5 (very severe). Lower scores indicate better health status. The percentage of participants with at least a 1-point improvement compared to baseline at Week 24 of Stage 2 in adult and pediatric (6-17 years of age) groups will be assessed
Stage 2: Percentage of participants with a radiological response at Week 24 of Stage 2 (pediatric participants 0-5 years of age) | Baseline, Week 24
  Radiological response defined by achieving at least 20% reduction in the sum of target lesion volumes (1 to 3 lesions), assessed by MRI by a BIRC at Week 24, provided that none of the individual target lesions has at least 20% increase from baseline and in absence of progression of non-target lesions and without new lesions. The percentage of participants with a radiological response at Week 24 of Stage 2 in pediatric participants 0-5 years of age will be assessed
Stage 2: Change from baseline in patient global impression of change (PGI-C) scale (adult and pediatric (6-17 years of age) participants) | Up to approximately 8 years
  PGI-C is a single item measure to assess the change in overall symptoms severity since the start of study. This single item instrument uses a 7-point rating scale, which ranges from 1 (very much improved) to 7 (very much worse). Lower scores indicate better health status. The change from baseline in PGI-C score will be assessed in adult and pediatric (6-17 years of age) participants
Stage 2: Change from baseline in patient-reported outcomes measurement information system (PROMIS) profile domains(adult and pediatric (6-17 years of age) participants) | Up to approximately 8 years
  The PROMIS-29 plus 2 Profile v2.1 (completed by adult participant) includes 29 items across domains of depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participant in social roles and activities, cognitive function abilities and pain intensity.
  The PROMIS Pediatric-25 Profile v2.0 (completed by children over 8 years of age) and PROMIS Parent-Proxy-25 Profile v2.0 (completed by parents for children under 8 years of age) include 25 items across the domains of depressive symptoms, anxiety, physical function-mobility, pain interference, fatigue, and peer relationships and pain intensity All items (except the pain intensity item) use a 5-point Likert scale, which ranges from 1 (not at all) to 5 (very much). The pain intensity item is scored on a 0-10 numeric rating scale, where 0 represents "no pain" and 10 represents "worst imaginable pain".
  The change from baseline in PROMIS domains will be assessed
Stage 2: Change from baseline in investigator global impression of change (IGIC) scale (adult and pediatric (6-17 years of age) participants) | Up to approximately 8 years
  The IGIC involves a single question that asks the investigator to rate the change in the patient's condition since the start of treatment or intervention, using a 7-point scale ranging from 1 (Very much improved) to 7 (Very much worse). The change from baseline in IGIC score will be assessed in adult and pediatric (6-17 years of age) participants
Stage 2: Change from baseline in health utilities of the EuroQol 5-dimension (EQ-5D) (adult and pediatric (6-17 years of age) participants) | Up to approximately 8 years
  The EQ-5D-5L (completed by adult participants) includes 5 items addressing dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with 5 response options, ranging from 1=no problems to 5=extreme problems The EQ-5D-Y (completed by children over 8 years of age) and EQ-5D-Y Proxy version (completed by parent for participants under 8 years of age or unable to record for themselves) includes 5 items addressing dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with 3 response options, ranging from 1= no problems to 3= a lot of problems
Stage 1 and 2: Duration of response (DOR) in adult and pediatric participants who receive alpelisib | Up to approximately 8 years
  DOR is defined as the time from first documented response until progression of LyM lesions by BIRC or death. This analysis only applies to participants who are on treatment with alpelisib (Stage 1 and 2) and who achieve response.
Stage 1: Radiological response rate of alpelisib in adult and pediatric (6-17 years of age) participants | Baseline, Week 24
  Radiological response defined by achieving at least 20% reduction in the sum of target lesion volumes (1 to 3 lesions), assessed by MRI by a BIRC at Week 24, provided that none of the individual target lesions has at least 20% increase from baseline and in absence of progression of non-target lesions and without new lesions.
  The percentage of participants (adult and pediatric 6-17 years of age) with radiological response at Week 24 of Stage 1 will be assessed.
Stage 1 and 2: Radiological response rate of alpelisib in adult and pediatric participants | Up to approximately 8 years
  Radiological response defined by achieving at least 20% reduction in the sum of target lesion volumes (1 to 3 lesions), assessed by MRI by a BIRC, provided that none of the individual target lesions has at least 20% increase from baseline and in absence of progression of non-target lesions and without new lesions.
  The percentage of participants who receive alpelisib (Stage 1 and 2) with radiological response will be assessed.
Stage 1 and 2: Alpelisib plasma concentrations | On Day 1 of Week 8, 16, 24, 48 and 120
  Alpelisib plasma concentrations in adult and pediatric participants (Stage 1 and 2).
Stage 1 and 2: Percentage of participants with of LyM-related symptoms, complications, and comorbidities on treatment with alpelisib in adult and pediatric participants at Week 24 | Week 24
  Percentage of participants with of LyM-related symptoms, complications, and comorbidities on treatment with alpelisib in adult and pediatric participants at Week 24 (Stage 1 and 2)
Stage 1 and 2: Percentage of participants with of LyM-related symptoms, complications, and comorbidities on treatment with alpelisib in adult and pediatric participants | Up to approximately 8 years
  Percentage of participants with of LyM-related symptoms, complications, and comorbidities on treatment with alpelisib in adult and pediatric participants (Stage 1 and 2)
Stage 1 and 2: Change from baseline in LyM lesions in adult and pediatric participants at Week 24 | Baseline, Week 24
  Change from baseline in the sum of target lesion volumes, the sum of MRI-measurable non-target lesion (if applicable) volumes, and the sum of all MRI-measurable lesion (target and non-target) volumes as assessed by BIRC at Week 24 in adult and pediatric participants (Stage 1 and 2)
Stage 1 and 2: Change from baseline in LyM lesions in adult and pediatric participants | Up to approximately 8 years
  Change from baseline in the sum of target lesion volumes, the sum of MRI-measurable non-target lesion (if applicable) volumes, and the sum of all MRI-measurable lesion (target and non-target) volumes as assessed by BIRC in adult and pediatric participants (Stage 1 and 2)
Stage 1 and 2: Percentage of participants with changes in non-target lesions in adult and pediatric participants at Week 24 | Baseline, Week 24
  Percentage of participants with changes in non-target lesions as assessed by BIRC at Week 24 in adult and pediatric participants (Stage 1 and 2)
Stage 1 and 2: Percentage of participants with changes in non-target lesions in adult and pediatric participants | Up to approximately 8 years
  Percentage of participants with changes in non-target lesions as assessed by BIRC in adult and pediatric participants (Stage 1 and 2)
Stage 1 and 2: Percentage of participants with new lesions in adult and pediatric participants at Week 24 | Baseline, Week 24
  The percentage of participants with new lesions as assessed by BIRC at Week 24 in adult and pediatric participants (Stage 1 and 2)
Stage 1 and 2: Percentage of participants with new lesions in adult and pediatric participants | Up to approximately 8 years
  The percentage of participants with new lesions as assessed by BIRC in adult and pediatric participants (Stage 1 and 2)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- United States (13):
  - UCSF Benioff Children s Hospital, Oakland, California
  - Lucile Packard Childrens Hosp, Palo Alto, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Childrens Hosp Boston Dept of Heme, Boston, Massachusetts
  - WA Uni School Of Med, St Louis, Missouri
  - Cinn Children Hosp Medical Center, Cincinnati, Ohio
  - Univ Hospital Of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health Science University, Portland, Oregon
  - CHOP Abramson Pediatric Resch Ctr, Philadelphia, Pennsylvania
  - Baylor College Of Medicine, Houston, Texas
  - U of TX Health Science Ct, Houston, Texas
  - Childrens Hospital and Regional Medical Center, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Brisbane, Queensland
- Novartis Investigative Site, Brussels, Belgium
- France (10):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
- Germany (5):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Berlin
- Italy (4):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Rotterdam, South Holland, Netherlands
- Spain (3):
  - Novartis Investigative Site, Esplugues, Barcelona
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com